CLINICAL TRIAL: NCT04223154
Title: The Effect of Dorsolateral Prefrontal Cortex Theta Burst Stimulation on Alcohol Cue Reactivity and Cognitive Control: a Double-blind, Sham Controlled Study of Heavy Alcohol Drinkers With a History of Alcohol Related Injury.
Brief Title: Effect of Theta Burst Stimulation on Alcohol Cue Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00063018
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder; Trauma Injury; Alcohol Dependence; Alcohol Abuse
Keywords: Transcranial Magnetic Stimulation; Brain Stimulation; Neuroimaging
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Accidental Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real TBS to the dlPFC (Experimental): One session of real intermittent Theta Burst Stimulation (TBS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC)
  Interventions: Device: Real iTBS to the dlPFC
- Sham TBS to the dlPFC (Sham Comparator): One session of sham Theta Burst Stimulation (TBS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC)
  Interventions: Device: Sham iTBS to the dlPFC

INTERVENTIONS:
Device: Real iTBS to the dlPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key).
  Arms: Real TBS to the dlPFC
Device: Sham iTBS to the dlPFC — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key).
  Arms: Sham TBS to the dlPFC

SUMMARY:
Alcohol Use Disorder (AUD) is prevalent, devastating, and difficult to treat. The intransigence of AUD is readily apparent in the Trauma Unit of Wake Forest University Baptist Hospital, wherein 23% of trauma related admissions are associated with alcohol - higher than the national average of 16%. Of these trauma related admissions, over 70% are estimated to have AUD and 41% will be likely be admitted to the trauma unit again within 5 years. While Dr. Veach (Co-Investigator) and her team in the Department of Surgery have demonstrated that a brief counseling intervention on the inpatient trauma unit can decrease morbidity and recidivism, the rates of AUD and relapse to drinking among these individuals remains very high. With a growing knowledge of the neural circuits that contribute to relapse in AUD, there is an emerging interest in developing a novel, neural-circuit specific therapeutic tool to enhance AUD treatment outcomes.

This will be achieved through a double-blind, sham-controlled cohort study in heavy alcohol drinkers with a history of alcohol-related injury. The brain reactivity to alcohol cues (Incentive Salience) and cognitive performance in the presence of an alcoholic beverage cue (Cognitive Control) will be measured immediately before and after participants receive real or sham intermittent theta burst stimulation (iTBS- a potentiating form of transcranial magnetic stimulation (TMS)) to the dorsolateral prefrontal cortex (dlPFC iTBS). The goals of this pilot study are to quantify the acute effect of a single session of real or sham dlPFC iTBS on brain response to alcohol cues (Aim 1) and cognitive flexibility in the presence of an alcohol cue (Aim 2) among risky drinkers (target engagement ).

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) is prevalent, devastating, and difficult to treat. The intransigence of AUD is readily apparent in the Trauma Unit of Wake Forest University Baptist Hospital, wherein 23% of trauma related admissions are associated with alcohol - higher than the national average of 16%. Of these trauma related admissions, over 70% are estimated to have AUD and 41% will be likely be admitted to the trauma unit again within 5 years. While Dr. Veach (Co-Investigator) and her team in the Department of Surgery have demonstrated that a brief counseling intervention on the inpatient trauma unit can decrease morbidity and recidivism, the rates of AUD and relapse to drinking among these individuals remains very high. With a growing knowledge of the neural circuits that contribute to relapse in AUD, there is an emerging interest in developing a novel, neural-circuit specific therapeutic tool to enhance AUD treatment outcomes. The long term goal of the multidisciplinary research team (Hanlon & Veach) is to develop an evidence-based brain stimulation treatment which can ultimately be prescribed to individuals that present to the Trauma Unit with AUD - decreasing their drinking and hospital recidivism.

The competing neurobehavioral decision systems (CNDS) theory posits that in addiction, choice results from a regulatory imbalance between two decision-making systems (impulsive and executive). These behavioral systems are functionally linked to two functional connectivity networks which regulate the incentive salience of the alcohol cue (Salience Network) and cognitive flexibility required for a vulnerable individual to shift attention away from the alcohol cue (Central Executive Network). Modulating these competing neural circuits (e.g. either dampening the incentive salience associated with alcohol cues (Strategy 1) or amplifying cognitive control in the presence of a cue (Strategy 2) may render alcohol users less vulnerable to relapse. Over the past 7 years, Dr. Hanlon's human brain stimulation research group has been focused on focused on Strategy 1 - dampening alcohol craving and brain reactivity to alcohol cues among heavy alcohol drinkers at risk for AUD or relapse to alcohol use. These studies led to a formal double-blind sham-controlled clinical trial of medial prefrontal cortex (mPFC) continuous theta burst stimulation (cTBS) in treatment-seeking alcohol users. Unfortunately, however, this approach is associated with more pain at the stimulation site (forehead) which undermines its promise as a tool to be readily scaled to a larger population, and it is not clear that this improves the attentional bias towards alcohol cues among these individuals.

Hence, the goal of this proposal is to evaluate Strategy 2 of the CNDS theory- increasing activity in executive control circuitry- as an innovative approach to dampening alcohol cue-reactivity (Aim 1) and improving cognitive control in the presence of an alcohol cue (Aim 2). This will be achieved through a double-blind, sham-controlled cohort study in heavy alcohol drinkers with a history of alcohol-related injury. The brain reactivity to alcohol cues (Incentive Salience) and cognitive performance in the presence of an alcoholic beverage cue (Cognitive Control) will be measured immediately before and after participants receive real or sham intermittent theta burst stimulation (iTBS- a potentiating form of transcranial magnetic stimulation (TMS)) to the dorsolateral prefrontal cortex (dlPFC iTBS). iTBS is a high-potency form of brain stimulation wherein two minutes of iTBS (600 pulses) leads to an increase in cortical excitability that lasts for approximately 30 minutes. In 2018 dlPFC iTBS was FDA-cleared as a treatment for major depressive disorder (wherein 30 sessions over 6 weeks lead to a sustained decrease in depressive symptoms for 6 months). In 2019, the first 2 manuscripts were published demonstrating that iTBS decreases cue-reactivity to cocaine. The goals of this pilot study are to quantify the acute effect of a single session of real or sham dlPFC iTBS on brain response to alcohol cues (Aim 1) and cognitive flexibility in the presence of an alcohol cue (Aim 2) among risky drinkers ("target engagement").

Aim 1: Evaluate the effect of dlPFC iTBS on alcohol cue-reactivity. The blood-oxygen level dependent (BOLD) signal associated with exposure to alcohol cues will be measured before and after sham and real iTBS using a validated, patient-tailored alcohol/non-alcoholic beverage cue task. Hypothesis: cue-evoked functional connectivity in the mPFC, anterior cingulate cortex (ACC), amygdala, and ventral striatum will be attenuated after real but not sham iTBS.

Aim 2: Evaluate the effect of dlPFC iTBS on cognitive performance in the presence of an alcohol cue. Following the alcohol cue reactivity task all individuals will perform the well-known alcohol Stroop task (downloaded from the NIH toolbox) on a Tablet PC while a glass of the participant's preferred alcoholic beverage (beer, wine, liquor) is placed within 5 feet of the participant (but out of arms length). This will occur before and after TBS. The participant will not be allowed to consume the drink. Hypothesis: Stroop accuracy and reaction time will be impaired at baseline, but this difference will be attenuated by real (but not sham) iTBS to the dlPFC (three way mixed model ANOVA, correcting for multiple comparisons).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-65.
2. Alcohol use disorder identification test score >7
3. Drink at least 20 standard sized alcohol beverage servings per week

Exclusion Criteria:

1. Current use of prescription or illicit psychoactive drugs (except marijuana or nicotine) known to decrease seizure threshold by self-report in the last 30 days.
2. Currently meets DSM-V criteria for substance use disorder for a substance other than alcohol, marijuana, or nicotine.
3. Has current suicidal or homicidal ideation.
4. Current breath alcohol concentration >0.002
5. Not currently at risk for withdrawal, as indicated by CIWA-Ar >5.
6. History of seizures or seizure disorder(s).
7. Females of childbearing potential who are pregnant (by urine HCG), planning to become pregnant, nursing, or who are not using a reliable form of birth control.
8. Any other violation of MRI/TMS safety measures.
9. Unable to read and understand questionnaires, assessments, and the informed consent.
10. No presence of metal objects in the head/neck.
11. History of traumatic brain injury resulting in hospitalization, loss of consciousness for more than 10 minutes, and/or having ever been informed he/she has an epidural, subdural, or subarachnoid hemorrhage.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Hanlon, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. All data is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real TBS to the dlPFC | Sham TBS to the dlPFC
Started | 8 | 3
Completed | 8 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | Real TBS to the dlPFC | Sham TBS to the dlPFC | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.2) | 40 (5.3) | 52 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
AUDIT score [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Use Disorders Identification Test (AUDIT) is a tool routinely used to assess the severity of alcohol use. It is scored on a scale of 0-40. The higher the AUDIT score, the more likely it is that the patient's drinking is affecting his/her health.
  units on a scale | 19.4 (6.6) | 21 (4) | 19.8 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Outcomes: Change in the k-Value, a Measure of Delay Discounting of Alcohol
Description: This outcome measure rates the change in k-value, or the delay discounting value of alcohol compared at baseline vs 1 hour after the intervention. Delay discounting is the tendency to place less value on rewards that are delayed in time. K typically falls between 0.0 and 0.5, with smaller values indicating a lack of discounting and a preference for delayed rewards, and higher values indicating stronger discounting and a preference for immediate rewards.
Time Frame: Baseline to 1 hour after the intervention
Population: Intent to treat population. There were no missing data.
Measure: Mean (Standard Deviation); unit: Change in k-value
Arm/Group | Real TBS to the dlPFC | Sham TBS to the dlPFC
Number analyzed (Participants) | 8 | 3
Change in k-value | -0.12 (0.27) | -7.42 (14.5)

2. Post Hoc Outcome: Neuroimaging Outcomes: Change in Brain Response to Alcohol Cues
Description: This will be measured using the blood oxygen level dependent signal in the prefrontal cortex
Time Frame: 1 hour after the intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Real TBS to the dlPFC | Sham TBS to the dlPFC
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT04223154/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04223154/ICF_001.pdf